CLINICAL TRIAL: NCT07387731
Title: Study of Fatigue and Respiratory Muscle Activation in the Spontaneous Breathing Test in Tube t Versus Support Ventilation at Mechanical Ventilation Weaning: Randomized Clinical Trial
Brief Title: Analysis on the Fatigue and Electromyographic Activation on the Mechanical Ventilation Weaning
Acronym: AFAEMG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Diogo Fanfa Bordin, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UFRGS_FAMED_EMG_D
Record Dates: First submitted 2017-05-07; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Electromyography; Ventilator Weaning; Critical Illness; Intensive Care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The binary randomization of the groups will be carried out through the electronic application Bracket RTSM (version 2.0.0, Global Bracket), and will be performed by a blind researcher to the groups evaluated.
  After evaluation of the eligibility criteria, the selected patients will be randomized into two groups: PSV Group (PSV) and T-tube group (TT), and will be cross-analyzed, with interval time between 30 minutes evaluations, the patient remaining In VM mode during this period.
Who Masked: Outcomes Assessor
Masking Description: Randomization, filtering of electromyographic data and statistical analysis will be performed by blind investigators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T tube method (Active Comparator)
  Interventions: Diagnostic Test: Sponteneous breathing test in T-tube
- Suport ventilation method (Active Comparator)
  Interventions: Diagnostic Test: Sponteneous breathing test in suport ventilation (PSV)

INTERVENTIONS:
Diagnostic Test: Sponteneous breathing test in T-tube — The intervention used in this study will be the two methods of weaning mechanical ventilation, T-tube and supportive ventilation already described in the arms of the study.
  Arms: T tube method
Diagnostic Test: Sponteneous breathing test in suport ventilation (PSV) — The intervention used in this study will be the two methods of weaning mechanical ventilation, T-tube and supportive ventilation already described in the arms of the study.
  Arms: Suport ventilation method

SUMMARY:
This study aims to evaluate respiratory muscle activation and fatigue during the mechanical ventilation weaning process using surface electromyography (sEMG). Despite various weaning methods, failure rates remain significant, necessitating objective evaluative tools. This randomized crossover clinical trial includes patients intubated for at least 24 hours who meet clinical criteria for a spontaneous breathing test (SBT). Participants will undergo two SBT methods: T-tube and Pressure Support Ventilation (PSV) at 7 cmH2O, each lasting 30 minutes and separated by a 30-minute washout period. Respiratory muscle activity will be quantified by the Root Mean Square (RMS) normalized to maximum inspiratory effort (%RMS), while muscle fatigue will be assessed through the Median Frequency (MF) of the power spectrum. The study seeks to determine which weaning method optimizes respiratory muscle performance and predicts extubation success, defined as 48 hours without ventilatory support.

DETAILED DESCRIPTION:
This randomized crossover clinical trial aims to compare the physiological effects of two spontaneous breathing trial (SBT) methods on respiratory muscle activity and fatigue in patients undergoing mechanical ventilation weaning. Patients intubated for at least 24 hours who meet clinical stability criteria-including adequate level of consciousness (Glasgow Coma Scale ≥ 13), hemodynamic stability without high doses of vasopressors, and an inspired oxygen fraction (FiO2) ≤ 0.4 - will be eligible for the study. Upon inclusion, participants will be randomized to one of two sequences: T-piece followed by Pressure Support Ventilation (PSV), or PSV followed by T-piece. The T-piece SBT involves disconnection from the ventilator with supplemental oxygen, while the PSV SBT is performed at 7 cmH2O with PEEP between 5-8 cmH2O. Each trial lasts 30 minutes, separated by a 30-minute washout period during which the patient is returned to their initial baseline ventilator settings to ensure physiological recovery and prevent carry-over effects. Electromyographic (sEMG) data will be captured using surface electrodes placed on the external intercostal muscles following SENIAM guidelines. Signal processing includes a Butterworth band-pass filter (20-450 Hz) and a sampling rate of at least 1000 Hz. The Root Mean Square (RMS) will be used to quantify muscle activation, normalized against the maximum inspiratory effort (%RMS) obtained during maximal inspiratory pressure (MIP) maneuvers. Muscle fatigue will be analyzed through the Median Frequency (MF) of the power spectrum using Fast Fourier Transform (FFT). Following the SBTs, patients will be extubated and monitored for 48 hours to determine the extubation success rate, defined as the absence of reintubation or rescue ventilatory support.Sample Size Calculation: The sample size was calculated based on the first five individuals evaluated, considering the mean and standard deviation of the primary outcome (%RMS) between the two evaluated methods. Adopting a significance level of 5% (a [alpha] = 0.05) and a statistical power of 80% (b [beta] = 0.80), the calculation indicated a required sample of [insira aqui o número total de pacientes, ex: 19] participants. To account for possible sample losses or technical signal artifacts, an additional 10% was added to the total.Statistical Analysis: Data distribution will be assessed using the Shapiro-Wilk test. Continuous variables will be expressed as mean and standard deviation or median and interquartile range, depending on normality. To compare the %RMS and MF between the T-piece and PSV methods, a Paired T-test or Wilcoxon Signed-Rank test will be utilized. For the analysis of time points (Baseline vs. 30th minute), a Two-way ANOVA for repeated measures with Post-hoc Bonferroni will be applied to identify significant differences and potential interaction effects between the weaning method and time. Categorical data, such as extubation success rate, will be analyzed using the Chi-square test or Fisher's Exact test. A p-value < 0.05 will be considered statistically significant for all analyses, which will be performed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

Patients will be intubated and ventilated mechanically for at least 24 hours, capable of starting the spontaneous breathing test based on the criteria recommended by the current Brazilian Recommendations on Mechanical Ventilation (Barbas, 2013), through a decision of the multiprofessional team. They should present adequate level of awareness to understand guidelines and age> 18 years.

-

Exclusion Criteria:

Patients with psychomotor agitation will not be able to interpret the electromyographic data, requiring an inspired fraction of oxygen greater than 0.6, tracheostomized, peritoniostomies and thoracotomies that would not allow the electrodes to be positioned in the right pectoralis major muscle, laparotomies that would not allow the positioning of the Electrodes in the rectus abdominis muscle and those whose family members have not adhered to the informed consent form (Appendix A).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Activation of Respiratory Muscles | Baseline, 30th minute of 1st Spontaneous Breathing Trial, 30th minute of washout (on initial mechanical ventilation settings), and 30th minute of 2nd Spontaneous Breathing Trial. Final minute of each phase used for analysis.
  Muscle activation of the respiratory muscles will be assessed using surface electromyography (sEMG). The raw signal will be processed to calculate the Root Mean Square (RMS), reflecting the magnitude of motor unit recruitment. To minimize inter-individual variability and allow for comparison across the crossover phases, all RMS values will be normalized as a percentage of the maximum inspiratory effort (MIE) recorded during a maximal inspiratory pressure (MIP) maneuver. Measurements will be recorded continuously during each phase of the trial: Baseline, the 1st Spontaneous Breathing Trial (SBT), the Washout period (on initial mechanical ventilation settings), and the 2nd SBT. For statistical analysis, the average value of the final minute of each specific phase will be used to compare the respiratory muscle load between different weaning modes.
Muscle Fatigue of Respiratory Muscles | Baseline, 30th minute of 1st Spontaneous Breathing Trial, 30th minute of washout (on initial mechanical ventilation settings), and 30th minute of 2nd Spontaneous Breathing Trial. Final minute of each phase used for analysis.
  Muscle fatigue will be evaluated through power spectrum analysis of the sEMG signal to determine the Median Frequency (MF). The MF is a sensitive physiological marker for detecting the early stages of myoelectric fatigue before clinical failure occurs. A significant downward shift in the MF from the beginning to the end of each study phase will be defined as an indicator of muscle fatigue. The assessment will follow the crossover protocol, collecting data at Baseline, during the 1st SBT, during the Washout period (to ensure return to muscular baseline), and during the 2nd SBT. Although data collection is continuous, the primary analysis will focus on the comparison of the MF values obtained in the final minute of each intervention phase to identify if one weaning strategy induces greater fatigue than the other.

SECONDARY OUTCOMES:
Clinical Tolerance to Extubation Success Rate within 48 hours | Patients are monitored continuously from the moment of endotracheal tube removal up to 48 hours post-extubation. Success or failure is definitively recorded at the 48-hour mark.
  Extubation success is defined as the patient's ability to maintain spontaneous breathing for a minimum of 48 hours following the removal of the endotracheal tube, without the need for reintubation or any form of rescue ventilatory support, including non-invasive ventilation (NIV). Clinical tolerance is monitored through standard weaning criteria, including a respiratory rate below 35 breaths per minute, oxygen saturation above 90% on FiO2 ≤ 40%, heart rate within 20% of baseline, and the absence of signs of increased respiratory work, such as accessory muscle use or paradoxical abdominal movement. The occurrence of reintubation or the necessity for ventilatory assistance within this 48-hour window is classified as extubation failure.

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Fanfa Bordin, Master, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided